CLINICAL TRIAL: NCT01364025
Title: Prophylactic Uterosacral Ligament Suspension at the Time of Hysterectomy for Prevention of Vaginal Vault Prolapse (PULS)
Brief Title: Prophylactic Uterosacral Ligament Suspension at the Time of Hysterectomy for Prevention of Vaginal Vault Prolapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaiser Permanente (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PULS
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Prolapse of Vaginal Vault After Hysterectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- uterosacral ligament suspension (Experimental): uterosacral ligament suspension colpopexy sutures will be placed bilaterally at the time of hysterectomy
  Interventions: Procedure: uterosacral ligament suspension colpopexy bilateral
- hysterectomy alone (No Intervention)

INTERVENTIONS:
Procedure: uterosacral ligament suspension colpopexy bilateral — Uterosacral ligament suspension colpopexy bilateral
  Other Names: uterosacral ligament suspension at the time of hysterectomy
  Arms: uterosacral ligament suspension

SUMMARY:
Is routine uterosacral ligament suspension an appropriate clinical adjunct at the time of hysterectomy?

The answers to these questions will facilitate the treatment of many American women. With the results of this study, the investigators would anticipate a reduction in the number of surgeries for pelvic organ prolapse. In addition, if uterosacral ligament suspension was shown to be ineffective, it would not be used routinely in the setting of hysterectomy and women will be spared the additional procedure and possibility of side effects or complications.

The relative risks and benefits of adding a prophylactic uterosacral ligament suspension at the time of hysterectomy in women without symptomatic prolapse symptoms have never been studied prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for primary procedure (hysterectomy either total or supracervical, performed either vaginally or abdominally, via laparoscopic or open approach)
* Eligibility for secondary procedure (uterosacral ligament suspension colpopexy)
* Prolapse in any compartment not extending beyond the hymen as measured by Pelvic Organ Prolapse Quantitative system
* No subjective complaints of Pelvic Organ Prolapse as determined by answer "no" to questions #3 of the short form of Pelvic Floor Distress Inventory: #3. Do you usually have a bulge or something falling out that you can see or feel in the vaginal area?

Exclusion Criteria:

* Contraindication for uterosacral ligament suspension colpopexy. (Surgeon's judgment that a contraindication to uterosacral ligament suspension colpopexy exists).
* Anticipated geographic relocation within the 12 months after surgery
* Inability to provide informed consent or to complete testing or data collection.

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2011-08; Primary Completion 2021-02-21 (Estimated); Study Completion 2021-02-21 (Estimated)

PRIMARY OUTCOMES:
To compare the occurrence of objective findings of pelvic organ prolapse beyond hymen after uterosacral ligament suspension of the vaginal apex at the time of hysterectomy vs. hysterectomy alone using Pelvic Floor Quantitative Examination | one year and annual thereafter for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Alperin, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente San Diego, San Diego, California, United States